CLINICAL TRIAL: NCT00087633
Title: A Randomized, Open-label Study of Prophylactic Administration of PEGASYS Plus Ribavirin After Liver Transplantation on Hepatitis C Recurrence in Patients With Hepatitis C
Brief Title: PHOENIX Study - A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) and COPEGUS (Ribavirin) Administered After Liver Transplantation for Hepatitis C.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18124
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: Copegus
- 2 (No Intervention)

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 135 micrograms subcutaneously (SC) weekly for 4 weeks followed by 180 micrograms SC weekly for 44 weeks
  Arms: 1
Drug: Copegus — 400 mg orally (PO) daily escalating to 1200 mg PO daily, for 48 weeks
  Arms: 1

SUMMARY:
This 2-arm study was designed to evaluate the efficacy, safety, and tolerability of prophylactic PEGASYS plus COPEGUS after liver transplantation for hepatitis C, compared to initiation of antiviral therapy at the time of clinical recurrence of hepatitis C infection. The anticipated time on study treatment was 3-12 months, and the target sample size was 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age
* Positive hepatitis C virus RNA at pre-transplantation
* Primary, single-organ recipient (cadaveric donor)
* Liver transplant between 10 and 16 weeks before treatment initiation

Exclusion Criteria:

* Multi-organ or re-transplant recipient
* Evidence of current hepatitis B infection
* Seropositive for human immunodeficiency (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (25):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Burlington, Massachusetts
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Newark, New Jersey
  - New York, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Madison, Wisconsin

REFERENCES:
- [Derived] Bzowej N, Nelson DR, Terrault NA, Everson GT, Teng LL, Prabhakar A, Charlton MR; PHOENIX Study Group. PHOENIX: A randomized controlled trial of peginterferon alfa-2a plus ribavirin as a prophylactic treatment after liver transplantation for hepatitis C virus. Liver Transpl. 2011 May;17(5):528-38. doi: 10.1002/lt.22271. PMID 21506241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 24 study centers in the US over a period of 4 years (12-Oct-04 - 17-Oct-08)
Pre-assignment Details: Eligible for the study were male or female patients ≥18 years of age with HCV infection who underwent orthotopic liver transplantation (OLT) because of liver cirrhosis attributed to HCV infection
Groups:
- Prophylaxis Arm: Pegylated interferon alfa-2a subcutaneously (SC) 135 μg/week for 4 weeks, then increased to 180 μg/week for the next 44 weeks, plus Ribavirin orally 400 mg/day (initial) to 1000 mg/day for patients <75 kg or 1200 mg/day for patients ≥75 kg PO (escalated) (maximum) administered orally
- Observation Arm: No antiviral therapy for HCV unless recurrence of HCV was histologically demonstrated. Once histological recurrence was demonstrated, patients received the same antiviral regimen as patients in the prophylaxis arm (ie, 48 weeks of combined PEG-IFN alfa-2a and ribavirin)
Period: Overall Study
Arm/Group | Prophylaxis Arm | Observation Arm
Started | 55 (Randomized) | 60 (Randomized)
Completed | 31 (Completed 48 weeks of treatment/observation) | 43 (Completed 48 weeks of treatment/observation)
Not Completed | 24 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylaxis Arm | Observation Arm | Total
Number analyzed (Participants) | 55 | 60 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (6.09) | 53.6 (5.37) | 52.5 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 45 | 48 | 93
Region of Enrollment [Number; unit: participants]
  United States | 55 | 60 | 115

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Histologically-confirmed Recurrence of Hepatitis C Virus (HCV)
Description: Histologically-confirmed recurrence of HCV defined as Batts-Ludwig inflammation grade ≥3 and/or fibrosis stage ≥2.
  Inflammation(Grade): 0 No Activity,1 Minimal,2 Mild,3 Moderate,4 Severe.
  Fibrosis (Stage): 0 No fibrosis, Normal; 1 Portal fibrosis; 2 Periportal fibrosis or rare portal septa; 3 Septal fibrosis, Fibrous septa with architectural distortion, no obvious cirrhosis; 4 Cirrhosis.
Time Frame: 120 weeks postrandomization
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Prophylaxis Arm | Observation Arm
Number analyzed (Participants) | 55 | 60
percentage of participants | 61.8 | 65.0
Statistical Analysis 1: Comparison: Prophylaxis Arm vs Observation Arm; Test type: Superiority or Other; p = 0.725, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-20.8 to 14.4]

2. Secondary Outcome: Summary of Virologic Response
Description: Rapid virologic responder (RVR): undetectable HCV-RNA at Week 4; complete early virologic responder (cEVR): undetectable HCV-RNA at Week 12; partial early virologic responder (pEVR): ≥2 log10 drop from baseline in HCV-RNA but positive at Week 12; early virologic responder (EVR): undetectable HCV-RNA or ≥2 log10 drop from baseline in HCV-RNA at Week 12; 24 weeks negative: undetectable HCV-RNA at Week 24; 48 weeks negative: undetectable HCV-RNA at Week 48; sustained virologic response (SVR): undetectable HCV-RNA at 24 weeks after the end of treatment.
Time Frame: After 4, 12, 24 and 48 weeks of therapy, and 24 weeks of follow-up
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Prophylaxis Arm | Observation Arm
Number analyzed (Participants) | 54 | 14
participants
  Rapid virologic responder (RVR) | 4 | 0
  Complete early virologic responder (cEVR) | 14 | 4
  Partial early virologic responder (pEVR) | 13 | 3
  Early virologic responder (EVR) | 27 | 7
  24 weeks negative | 20 | 6
  48 weeks negative | 18 | 3
  Sustained virologic responder (SVR) | 12 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the period of the study (4 years, 12-Oct-2004 - 17-Oct-2008)
Description: Safety Population: 54 patients in the prophylaxis arm, and 60 patients in the observation arm. One patient randomized to the prophylaxis arm was excluded from the safety population because they withdrew consent before receiving any study medication and did not have any postbaseline assessments.
Arm/Group | Prophylaxis Arm | Observation Arm
Serious Adverse Events (participants affected / at risk) | 25/54 | 21/60
Other Adverse Events (participants affected / at risk) | 54/54 | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis Arm (N=54) | Observation Arm (N=60)
Infections and infestations (Infections and infestations) | 6 (7) | 6 (8)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (8) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 6 (6) | 3 (3)
Blood and lymphatic system disordersimag (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Cardiac disorders (Cardiac disorders) | 0 (0) | 2 (2)
Investigations (Investigations) | 2 (2) | 0 (0)
Surgical and medical proceduresi (Surgical and medical procedures) | 0 (0) | 2 (2)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0)
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions (General disorders) | 5 (5) | 1 (1)
Injury, poisoning and procedural complicationsE (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Nervous system disorders (Nervous system disorders) | 4 (4) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 3 (3) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis Arm (N=54) | Observation Arm (N=60)
General Disorders and administration site conditions (General disorders) | 48 (108) | 33 (62)
Gastrointestinal disorders (Gastrointestinal disorders) | 44 (114) | 37 (84)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 43 (79) | 17 (20)
Nervous system disorders (Nervous system disorders) | 41 (76) | 25 (43)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 31 (60) | 27 (43)
Psychiatric disorders (Psychiatric disorders) | 30 (44) | 17 (25)
Infections and infestations (Infections and infestations) | 26 (35) | 24 (41)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 25 (47) | 23 (33)
Investigations (Investigations) | 24 (37) | 29 (52)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 23 (31) | 15 (27)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 21 (32) | 14 (19)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 16 (21) | 17 (24)
Renal and urinary disorders (Renal and urinary disorders) | 13 (17) | 13 (16)
Vascular disorders (Vascular disorders) | 13 (15) | 13 (15)
Eye disorders (Eye disorders) | 10 (14) | 6 (7)
Hepatobiliary disorders (Hepatobiliary disorders) | 9 (12) | 8 (15)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 8 (9) | 3 (3)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 5 (5)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 (2) | 4 (5)
Cardiac disorders (Cardiac disorders) | 3 (3) | 3 (3)
Endocrine disorders (Endocrine disorders) | 2 (2) | 3 (3)
Social circumstances (Social circumstances) | 1 (1) | 0 (0)
Immune system disorders (Immune system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.